CLINICAL TRIAL: NCT02482324
Title: A Phase I, Randomized, Open-Labeled Pharmacokinetic Study of ALZT-OP1 in Normal Healthy Volunteers
Brief Title: Phase 1 Study of ALZT-OP1 Combination Therapy in Normal Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AZTherapies, Inc. (Industry)
Collaborators: Panax Clinical Research (Other); Pharma Consulting Group AB (Industry); KCAS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AZT-002
Record Dates: First submitted 2015-06-22; First posted 2015-06-26 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Cromolyn Sodium; Ibuprofen; Dry Powder Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A-B (Other): 12 subjects will receive a single oral inhaled dose of ALZT-OP1a, via dry powder inhaler, and a single oral tablet dose of ALZT-OP1b on Day 1, and two doses of ALZT-OP1a and ALZT-OP1b on Day 2, within two minutes of each other. All subjects will have plasma collected for PK analysis and 6 of 12 consented subjects from this group will provide CSF samples for analysis. CSF collected on Day 1 only.
  Interventions: Drug: ALZT-OP1a; Drug: ALZT-OP1b; Device: Dry Powder Inhaler
- Treatment B-A (Other): 12 subjects will receive two oral inhaled doses of ALZT-OP1a, via dry powder inhaler, and two oral tablet doses of ALZT-OPb, within two minutes of each other, on Day 1, and single doses of ALZT-OP1a and ALZT-OP1b on Day 2. All subjects will have plasma collected for PK analysis and 6 of 12 consented subjects from this group will provide CSF samples for analysis. CSF collected on Day 1 only.
  Interventions: Drug: ALZT-OP1a; Drug: ALZT-OP1b; Device: Dry Powder Inhaler

INTERVENTIONS:
Drug: ALZT-OP1a — Mast cell stabilizer
  Other Names: Cromolyn, Intal
Drug: ALZT-OP1b — anti-inflammatory
  Other Names: ibuprofen
Device: Dry Powder Inhaler — The inhaler will be used to deliver ALZT-OP1a via oral inhalation for both days on study.

SUMMARY:
This is an open-labeled, cross-over design, pharmacokinetic study, to determine the pharmacokinetics of ALZT-OP1 (a combination drug therapy) designated as ALZT-OP1a and ALZT-OP1b, in both plasma and CSF, following co-administration of the active compounds, in healthy volunteers, aged 55-75, and in good general health.

DETAILED DESCRIPTION:
This is an open-labeled, cross-over design, pharmacokinetic study, where 24 subjects will be randomly assigned to receive treatment regimen A-B or B-A on two consecutive days of dosing.

Two dosing groups are planned for the study :

* Group 1 (n=12)
* Group 2 (n=12)

Each group will be admitted to the Phase I Unit the evening before dosing and will initiate dosing the next morning for 2-days of consecutive treatment (A-B, or B-A). Both groups will undergo identical study related procedures, except those subjects that consent to CSF collection on Day 1 of dosing.

Dose regimen A consists of a single inhaled oral dose of ALZT-OP1a via dry powder inhaler + a single oral tablet dose of ALZT-OP1b.

Dose regimen B consists of two oral inhaled doses of ALZT-OP1a, not more than 2 minutes apart, via dry powder inhaler + two oral tablet doses of ALZT-OP1b.

Plasma Collection, All Subjects (n=24) 1 mL blood samples will be collected at T: 0, 5, 10, 15, 30, 1 hr, 2 hr, 4 hr, and 6 hours, following ALZT-OP1 administration (Days 1 and 2).

CSF Collection, Sub-group (n=12) A sub-group of 12 subjects will be consented for CSF collection.

1 mL of CSF will be collected at T: 0, 5 min, 30 min, 2 hr, and 4 hours, following ALZT-OP1 administration (Day 1 only).

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed written informed consent;
* Age 55-75 inclusive;
* ECG within normal limits;
* Body mass index (BMI) ≥ 18 kg/m2 and ≤ 30 kg/m2;
* Negative urine drug screen for selected drugs of abuse at screening;
* Negative for hepatitis and HIV at screening;
* Good general health, as determined by medical history, physical examination, and clinical laboratory testing;
* Willingness to stay in the unit overnight for the duration of the study;
* Consent for CSF collection (for those in CSF group).

Exclusion Criteria:

* Current smokers, or ex-smokers with a remote history (> 100 pack/year);
* Clinically significant medical conditions;
* History of ECG abnormalities;
* Symptomatic viral infection, or suspicion thereof (including rhinitis) in the last 14 days prior to dosing;
* Signs of active pulmonary infection or other pulmonary inflammatory conditions, even in absence of febrile episodes, in the last 14 days;
* History or presence of disease in the kidneys and/or heart, lungs, liver, gastrointestinal tract, endocrine organs or other conditions such as metabolic disease known to interfere with the absorption, distribution, metabolism, and excretion of drugs;
* Malignancy, regardless of location;
* Autoimmune disorders such as (but not limited to) lupus erythematosus, multiple sclerosis, rheumatoid arthritis, or sarcoidosis;
* Investigational agents are prohibited one month prior to entry and for the duration of the trial;
* Currently taking medications known to be CYP2C9 inducers (i.e. carbamazepine and rifampicin);
* Currently taking cromolyn, or have taken cromolyn, within the past 30 days;
* NSAID use (products containing ibuprofen while on study);
* Aspirin, or products containing aspirin, while on study;
* Allergy or hypersensitivity to cromolyn (also known as Intal®, Nasalcrom®, etc.);
* Allergy or hypersensitivity to ibuprofen (Advil®, Motrin®, Nuprin®, etc.) or aspirin, including Stevens-Johnson syndrome;
* History of hypersensitivity or allergies to any of the drug compound under investigation (cromolyn, ibuprofen, lactose, or magnesium stearate);
* History of clinically significant respiratory disorders and chronic respiratory disease with impaired respiratory effort or difficulty taking inhaled drugs (examples: COPD, emphysema);
* Abnormal pulmonary function test, defined for this protocol as: FEV1/FVC < 70% of the predicted value for the subject, when compared to reference values; AND FEV1 and FVC < 70% of predicted value when compared to reference values, indicating moderate to severe respiratory obstruction;
* Any other disease or condition, which, in the opinion of the investigator, would make the subject unsuitable for this study;
* Female subjects of reproductive potential with a positive pregnancy test (urine or serum) or who are pregnant or lactating.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-06; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Non-compartmental plasma pharmacokinetics for ALZT-OP1a and ALZT-OP1b | T=0 to 6 hours (0, 5, 10, 15, 30, 60, 120, 240, and 360 minutes)
  * AUC (0-∞) (area under the curve from 0 to infinity)
  * AUC (0-t) (area under the curve from 0 to t hours where t is the last measured concentration
  * AUCPLASMA/AUCCSF (ratio at 5 min, 30 min, 2 hr and 4 hours)
  * CL/F (apparent total body clearance)
  * Cmax (maximum plasma concentration observed)
  * T ½ (half life)
  * Tmax (sampling time at which Cmax occurred)
  * Vd/F (apparent volume of distribution
  Plasma concentration-time profiles will be presented for both study drugs.

SECONDARY OUTCOMES:
Levels of ALZT-OP1a and ALZT-OP1b in cerebrospinal fluid (CSF) | T=0 to 4 hours (0, 5, 30, 120, and 240 minutes)
  CSF samples will be collected at 5 time-points to measure levels of ALZT-OP1a and ALZT-OP1b in CSF.
Number of Treatment Emergent Adverse Events (TEAE) | 2 days
  Safety will be evaluated based on the number, type, and frequency of treatment emergent adverse events. They will be individually presented for all subjects in data listings, and summarized in tables by treatment group and by treatment assignment. The AEs will be summarized and reported collectively based on information obtained through physical examination, ECG, and laboratory findings captured after dosing was initiated.

CONTACTS AND LOCATIONS:
Overall Officials: David Elmaleh, PhD, Study Chair — Study Sponsor; David Brazier, BS, Study Director — Study Sponsor
Locations (1):
- Panax Clinical Research, Miami Lakes, Florida, United States